CLINICAL TRIAL: NCT04251195
Title: Verbal Memory Training Using Virtual Reality in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Ottawa Mental Health Centre (Other)
Responsible Party: Principal Investigator, Synthia Guimond, Scientist, The Royal Ottawa Mental Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018048
Record Dates: First submitted 2020-01-27; First posted 2020-01-31 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Intervention (Experimental)
  Interventions: Behavioral: Cognitive Intervention
- Active Control Intervention (Active Comparator)
  Interventions: Behavioral: Active Control Intervention

INTERVENTIONS:
Behavioral: Cognitive Intervention — Participants will undergo 15 minutes of a cognitively challenging activity in the Virtual Reality environment. (More details about each condition will be added after study completion to protect the blinding of our participants).
  Arms: Cognitive Intervention
Behavioral: Active Control Intervention — Participants will undergo 15 minutes of a cognitively challenging activity in the Virtual Reality environment. (More details about each condition will be added after study completion to protect the blinding of our participants).
  Arms: Active Control Intervention

SUMMARY:
Verbal episodic memory is an independent declarative memory system associated with language and is responsible for storage and conscious recall of previous personal experiences. Verbal episodic memory is impaired in schizophrenia and is related to patients' functional outcomes. Because no medication has shown clear positive effects on verbal memory impairment in schizophrenia, there is a great need to find effective cognitive remediation treatments (CRT) that could improve this domain in this psychiatric population. Although CRT programs have shown small to moderate positive effects on verbal memory in individuals with schizophrenia, traditional lab-based computerised cognitive interventions have notable attrition rates. In recent years, along with the advancement of technology, the development of Virtual Reality (VR) has allowed the possibility for new training techniques. Previous studies have established the initial feasibility and safety of using VR in schizophrenia population. However, no studies have examined the feasibility, safety and efficacy of combining VR technology with verbal memory training among individuals with schizophrenia. Thus, in this study, we will adapt an exercise from the Strategy for Semantic Association Memory (SESAME; (Guimond et al., 2018; Guimond & Lepage, 2016) training to a VR environment. We aim to determine the feasibility of using virtual reality in the context of a cognitive remediation intervention and to assess the initial efficacy of our verbal memory training on the use of semantic encoding strategies in people with schizophrenia. We also aim to assess participants' experience and tolerability of the VR training.

DETAILED DESCRIPTION:
In this study, participants will first undergo the Hopkins Verbal Learning Test - Revisited (HVLT-R) to assess the baseline use of semantic clustering and verbal memory recall performance. Participants will then be randomly assigned to either a control group or a verbal training group. Participants in both groups will undergo a short session (15 minutes) of VR training. Finally, participants will be invited to perform an alternate version of the HVLT-R to assess initial change in semantic clustering and verbal memory recall performance after the training. They will also complete the VR Experience Questionnaire and the simulator sickness questionnaire (SSQ) in order for the research team to gain feedback from participants regarding their experience and tolerability of the VR session.

ELIGIBILITY:
Inclusion Criteria:

* age 20-60 years
* the ability to read and speak fluent English
* having a diagnosis of schizophrenia or schizoaffective from a psychiatrist and confirmed by the Mini International Neuropsychiatric Interview (M.I.N.I) interview
* considered clinically stable (on stable medication for more than one month, and have a score below 95 on the Positive and Negative Syndrome Scale (PANSS))

Exclusion Criteria:

* having vision problems that cannot be corrected with contact lenses or glasses that fit into the VR goggles (because of requirements of VR headset)
* having significant neurological or medical disorders (other than schizophrenia/schizoaffective disorder) that may produce cognitive impairment
* a recent history of substance abuse or dependence (within the past 3 months)
* decisional incapacity requiring a guardian
* having past or current conditions of seizure, epilepsy, migraines or cybersickness

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Change in semantic encoding strategy use as measured by change in semantic clustering from baseline - the Hopkins Verbal Learning Test - Revisited (HVLT-R). | baseline, post treatment (~20 minutes)
  The Hopkins Verbal Learning Test - Revisited (HVLT-R) for verbal memory is a 12-item test to measure a person's ability to encode, combine, store and recover verbal information in memory.
Feasibility of the intervention | baseline, post treatment (~20 minutes)
  Feasibility of the intervention as measured by the number of people who complete the intervention.

SECONDARY OUTCOMES:
Change in verbal memory performance from baseline | baseline, post treatment (~20 minutes)
  The Hopkins Verbal Learning Test - Revisited (HVLT-R) for verbal memory is a 12-item test to measure a person's ability to encode, combine, store and recover verbal information in memory.
Participants' experience and tolerability - VR experience questionnaire | post treatment (~20 minutes)
  VR experience questionnaire is a 5-item questionnaire that our research team designed to obtain feedback from participants regarding their experience with the VR intervention following the completion of the VR session.
Participants' experience - Simulator sickness questionnaire (SSQ) | post treatment (~20 minutes)
  Simulator sickness questionnaire (SSQ) is a 16-item questionnaire developed to examine the degree of cybersickness in participants after the use of VR.

CONTACTS AND LOCATIONS:
Overall Officials: Synthia Guimond, PhD, Principal Investigator — Royal Ottawa Mental Health Center
Locations (1):
- Royal Ottawa Mental Health Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data collected from this study may be shared with other researchers at the Royal's Institute of Mental Health Research for analyses and re-analyses. Variables of the study and scripts used for analyses will be made available to the public. De-identified data will also be shared with the general public upon request. Data that can connect with participants' identity will NOT be used or shared for analyses.
Supporting Information: SAP, Analytic Code
Time Frame: De-identified data will become available upon completion of the study and once results have been published in an academic journal (anticipated time frame: the year of 2021).

REFERENCES:
- [Result] Guimond S, Lepage M. Cognitive training of self-initiation of semantic encoding strategies in schizophrenia: A pilot study. Neuropsychol Rehabil. 2016;26(3):464-79. doi: 10.1080/09602011.2015.1045526. Epub 2015 Jul 6. PMID 26145159
- [Result] Guimond S, Beland S, Lepage M. Strategy for Semantic Association Memory (SESAME) training: Effects on brain functioning in schizophrenia. Psychiatry Res Neuroimaging. 2018 Jan 30;271:50-58. doi: 10.1016/j.pscychresns.2017.10.010. Epub 2017 Oct 25. PMID 29102504